CLINICAL TRIAL: NCT01133886
Title: Use of Decitabine in Myelodysplastic Syndrome (MDS) Following Azacitidine (AZA) Failure
Acronym: DEC-MDS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: King's College London (Other)
Collaborators: King's College Hospital NHS Trust (Other)
Responsible Party: Professor Ghulam Mufti, King's College London
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DEC-MDS
Record Dates: First submitted 2010-05-28; First posted 2010-05-31 (Estimated); Last update posted 2010-09-03 (Estimated); Status verified 2010-09

CONDITIONS: Acute Myeloid Leukemia; Chronic Myelomonocytic Leukemia; Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Chronic; Myelodysplastic Syndromes | interventions — Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Decitabine (Experimental)
  Interventions: Drug: Decitabine

INTERVENTIONS:
Drug: Decitabine — Patients will receive decitabine as a 20mg/m2 one hour intravenous infusion once daily on days 1 to 5 of a 4 week cycle.
  Other Names: Dacogen

SUMMARY:
The purpose of this study is to assess the response rate at 6 months in Myelodysplastic Syndrome (MDS) patients, Chronic Myelomonocytic Leukaemia (CMML-2) patients, and Acute Myeloid Leukaemia (AML) patients with up to 30% bone marrow blasts, treated with low-dose decitabine who have previously failed therapy with 5-azacitidine.

ELIGIBILITY:
Inclusion Criteria:

1. Written signed informed consent.
2. ≥18 years of age.
3. Diagnosed MDS with 5% or more marrow blasts and IPSS risk intermediate 2 or high risk; or chronic myelomonocytic leukemia (CMML-2); or AML with 20-30% bone marrow blasts.
4. Patients who have failed therapy with azacitidine.
5. Performance status 0-2 (ECOG scale).
6. Adequate hepatic (bilirubin < 1.5 X ULN or AST< 2.5 X ULN) and renal functions (creatinine <1.5 X ULN).

Exclusion Criteria:

1. Nursing and pregnant females.
2. Females of childbearing potential and males not willing to practice an effective method of contraception whilst receiving decitabine and for 2 months after the last infusion.
3. Patients with previous malignancy or concurrent malignancy.
4. Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure and unstable angina pectoris.
5. Ongoing oral corticosteroids are not permitted. However, use of corticosteroids (topical and inhaled) is permitted and prophylactic steroids are allowed for transfusion reactions.
6. Patients who have received any investigational agent within the 30 days preceding the first dose of study drug.
7. Patients who have received prior intensive combination chemotherapy or high-dose cytarabine (>/= 1g/m*2 per dose). (Prior biologic therapies, targeted therapies and single agent chemotherapy are allowed).
8. Patients who have an active viral or bacterial infection. Note: No patient is allowed to enter the study unless infections have been fully treated and the patient has remained afebrile for 7 days without antibiotics.
9. Patients who have concurrent autoimmune hemolytic anemia or immune thrombocytopenia.
10. Patients who have previously been treated with decitabine.
11. Patients who have known positive serology for HIV.
12. Patients with a condition that may be unable to comply with the treatment and monitoring requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-09; Primary Completion 2012-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Overall response rate in the efficacy-evaluable (EE) population | 6 months

SECONDARY OUTCOMES:
Overall survival | 18 months
Time to AML progression (for MDS and CMML-2 patients only) or death | 18 months
Haematological improvement | 18 months
Transfusion requirements | 18 months
Cytogenetic response | 18 months
Treatment related toxicity | Up until one month after last IMP dose

CONTACTS AND LOCATIONS:
Overall Officials: Ghulam J Mufti, MB, DM, FRCP, FRCPath, Principal Investigator — King's College London
Locations (1):
- King's College Hospital NHS Foundation Trust, London, United Kingdom